CLINICAL TRIAL: NCT02964988
Title: uPAR PET/CT in Radium-223-dichloride Treatment of Patients With Metastatic Castration-resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issues and interim results
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Marie Øbro Fosbøl, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK-2016-PC-1; 2016-002184-34 (EudraCT Number)
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer Metastatic; Bone Metastases
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- uPAR PET/CT (Experimental): Injection of 68Ga-NOTA-AE105 followed by PET/CT scan. Administration will be performed twice in approximately 8 weeks.
  Interventions: Drug: Injection of PET tracer 68Ga-NOTA-AE105; Device: PET/CT

INTERVENTIONS:
Drug: Injection of PET tracer 68Ga-NOTA-AE105 — Following injection of 68Ga-NOTA-AE105 the patients will be subjected to whole body PET/CT
Device: PET/CT — Whole body PET/CT

SUMMARY:
The purpose of this study is to investigate the applicability of urokinase plasminogen activator receptor (uPAR) Positron Emission Tomography (PET) / CT molecular imaging in patients with metastatic castration-resistant prostate cancer (mCRPC)

DETAILED DESCRIPTION:
68Ga-NOTA-AE105 is a radioligand targeting urokinase plasminogen activator receptor (uPAR), which is a promising imaging biomarker of tumor aggressiveness. 68Ga-NOTA-AE105 PET/CT will be applied in patients with mCRPC during treatment with Radium-223. PET/CT will be performed before initiation of Radium therapy and after two treatment cycles. The initial semiquantitative uptake (standard uptake values, SUVs) of 68Ga-NOTA-AE105 in metastases as well as the change in these parameters after therapy will be correlated with overall survival and progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration resistant prostate cancer
* Approved to receive Radium-223 therapy
* Written and oral consent

Exclusion Criteria:

* Lack of communication skills
* Other known malignant disease
* Known allergy towards IMP
* Severe claustrophobia
* If a participant exhibits allergic reaction i the IMP, the participant will be excluded from further participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01; Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
uPAR PET/CT imaging | 1 hour post injection
  Standard uptake values (SUVs) of 68Ga-NOTA-AE105 evaluated on uPAR-PET/CT scan performed within 1 hour following injection of 68Ga-NOTA-AE105
Change in uPAR PET/CT after two cycles of Radium-223 | 8 weeks
  Change in Standard uptake values (SUVs) of 68Ga-NOTA-AE105 evaluated on uPAR-PET/CT scan performed after 2 cycles of Radium-223 therapy

SECONDARY OUTCOMES:
uPAR PET/CT as prognostic factor for overall survival | 12 months
  Patients will be followed for 12 months after uPAR PET/CT
uPAR PET/CT as prognostic factor for progression free survival | 12 months
  Patients will be followed for 12 months after uPAR PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fosboel, MD, Principal Investigator — Rigshospitalet, Department of Clinical Physiology, Nuclear Medicine & PET
Locations (1):
- Rigshospitalet, Copenhagen, Denmark